CLINICAL TRIAL: NCT04890015
Title: The Impact of Transanal Decompression Tube Placement on Anastomotic Dehiscence After Colorectal Anastomosis. A Randomized and Controlled Clinical Trial
Brief Title: The Impact of Transanal Decompression Tube Placement After Colorectal Anastomosis: A Randomized Trial
Acronym: SONDES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta (Other)
Responsible Party: Principal Investigator, Ander Timoteo Delgado, General and digestive surgeon, Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 62019
Record Dates: First submitted 2021-05-12; First posted 2021-05-18 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Colorectal Cancer; Postoperative Complications; Anastomotic Leak; Anastomotic Complication
Keywords: Colorectal cancer; Transanal tube emplacement; Anastomotic leakage
MeSH Terms: conditions — Colorectal Neoplasms; Postoperative Complications; Anastomotic Leak

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intraoperative transanal decompression tube placement (Experimental): Intraoperatively under direct vision in the lower rectum, the balloon of the catheter will be inflated with 5-10cc of distilled water and it will be secured with a dressing / tape to the buttock connected to a collection bag.
  Interventions: Procedure: Intraoperative transanal decompression tube placement
- Non intraoperative transanal decompression tube placement (No Intervention): The usual postoperative care approved by the unit will be followed.

INTERVENTIONS:
Procedure: Intraoperative transanal decompression tube placement — Intraoperatively under direct vision in the lower rectum, the balloon of the catheter will be inflated with 5-10cc of distilled water and it will be secured with a dressing / tape to the buttock connected to a collection bag.
  Arms: Intraoperative transanal decompression tube placement

SUMMARY:
There is currently no standardization in the use of the transanal decompressive tube during the postoperative after a colorectal surgery. The available evidence is based on studies with methodological differences. Most of the studies exclude patients with a diverting ileostomy, which are those patients who have a higher risk of anastomotic leak, so the real effect of transanal decompressive tube could have been masked. For this reason we believe that to assess the true effect of rectal decompression, patients with diverting stoma should be included.

DETAILED DESCRIPTION:
One of the complications of performing the colorectal anastomosis is the anastomotic leak, which sometimes entails the need for reinterventions and stoma formation (provisional or definitive). In recent decades, the improvement in surgical techniques together with the knowledge of the causes that predispose to the anastomotic failure have allowed to reduced the rates.

The placement of a tube probe through the anus in the postoperative period that decompresses the contents of the interior of the intestine (liquid or air) has been proposed as a factor that could influence the healing between intestines.

In studies carried out in other centers, with the same characteristics as the present one, differences have been shown in the probability of anastomotic leakage, but these results are not conclusive and do not allow us to know the effectiveness of this procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing scheduled laparoscopic, robotic or laparotomic colorectal cancer surgery who undergo colorectal anastomosis.
* Both mechanical and manual colorectal anastomosis with or without diverting ileostomy.
* Negative intraoperative air-leak test.
* Height of the anastomosis: promontory or distal to it.
* Age≥18 years.
* Histology of Adenocarcinoma with or without prior neoadjuvant treatment.
* Any T, any N, any M.
* Informed consent signed by the patient and by the researcher.

Exclusion Criteria:

* No performance of colorectal anastomosis.
* Colorectal tumor with histology other than adenocarcinoma or adenoma.
* Patients with psychiatric illnesses, addictions or any disorder that prevents understanding of surgery.
* Inability to read or understand any of the informed consent languages (Catalan, Spanish).
* Emergency surgery.
* Any patient who, due to his medical characteristics, presents a high individual risk when being included and completing the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2017-07-10 (Actual); Primary Completion 2023-06-10 (Estimated); Study Completion 2023-07-10 (Estimated)

PRIMARY OUTCOMES:
Anastomotic leakage rate between treatment arms | Within 30 days after surgery
  Anastomotic leakage (No/Yes), degree of anastomotic leakage (A, B or C), days of anastomotic leak diagnosis after colorectal surgery

SECONDARY OUTCOMES:
Reintervention rate | Within 30 days after surgery
  Reintervention due to any cause within 30 days after surgery
Postoperative complication rate | Within 30 days after surgery
  Rate of medical and surgical complications within 30 days after surgery using the Dindo-Clavien classification, described as:
  Grade I = Any deviation from the normal postoperative course. Grade 2 = Requiring pharmacological treatment with drugs other than such allowed for grade I complications.
  Grade III = Requiring surgical, endoscopic or radiological intervention, not under (Grade IIIa) or under general anesthesia (Grade IIIb) Grade IV = Life-threatening complication with single organ (Grade IVa) or Multiorgan dysfunction (Grade IVb) Grade V = Death of a patient.
Definitive and / or temporary stoma rate after anastomotic leakage | Within 30 days after surgery
  Stoma formation due to anastomotic leak (No/Yes)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Dr. Josep Trueta de Girona, Girona, Spain